CLINICAL TRIAL: NCT00240513
Title: A Randomized Study to Compare the Acne Relapse Rate After a 3-mo Course of Oral Minocycline, to a 3-mo Course of Oral Minocycline in Combination With a Daily Dose of Topical Tretinoin 0.01% Followed by 3 mo of Topical Tretinoin Alone
Brief Title: Study Comparing Acne in Patients Taking Oral Minocycline to Patients Taking Minocycline Plus Topical Tretinoin
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Too much difficulty recruiting and retaining patients, PI decided to stop.
Sponsor: Derm Research @ 888 Inc. (Industry)
Collaborators: Stiefel, a GSK Company (Industry)
Responsible Party: Principal Investigator, David Richard THOMAS, MD FRCP(C), Derm Research @ 888 Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2004-03
Record Dates: First submitted 2005-10-16; First posted 2005-10-18 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Acne Vulgaris
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Minocycline; Tretinoin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minocycline 3 mo (Active Comparator): Minocycline 3 mo
  Interventions: Drug: Minocycline
- Minocycline plus Tretinoin (Experimental): Minocycline plus Tretinoin for 3 months
  Interventions: Drug: Minocycline plus tretinoin

INTERVENTIONS:
Drug: Minocycline — 100 mg capsules OD for 3 months
  Other Names: Minocin
  Arms: Minocycline 3 mo
Drug: Minocycline plus tretinoin — 100mg OD Minocycline for 12 weeks plus OD Topical tretinoin 0.01% for 12 weeks Followed by topical tretinoin 0.01% OD for 12 weeks alone
  Other Names: Minocin; Tretinoin
  Arms: Minocycline plus Tretinoin

SUMMARY:
The use of oral antibiotics alone to treat inflammatory acne provides little to no long term therapeutic benefit.

Acne relapse rates can be reduced by using topical tretinoin 0.01% in conjunction with minocycline, thereby increasing the therapeutic effect of the oral antibiotic.

DETAILED DESCRIPTION:
Although oral antibiotics have been the mainstay of treatment of inflammatory acne for 30 years, studies comparing their efficacy have little scientific value.

Evidence-based dermatology proves minocycline to be an effective treatment for acne vulgaris while the patient remains on the medication; however, the relapse rate of acne after a course of antibiotics has never been established.

The relapse rate would appear to be significant, as repeated courses and long-term antibiotic use are commonly prescribed in practice. The increasing problem of drug resistance has raised issues of the suitability of such long term antibiotic treatment and this overuse is probably a contributing factor of multiple drug resistance in our society.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written consent
* Either sex
* Any age
* Diagnosis of acne vulgaris with a minimum of 20 inflammatory acne lesions on the face.

Exclusion Criteria:

* Known hypersensitivity to tetracyclines
* Use of any oral antibiotics in the previous 3 months
* Pregnancy, breast-feeding or lactating
* Inability or unwillingness to comply with the requirements of the protocol, or agree to the use of their data as determined by the investigator.
* Concomitant medical condition which, in the investigator's opinion, may confound the study results or interfere with study assessments or outcomes.
* Patients with severe acne on the chest, back or trunk.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Long-term efficacy | 4 years

SECONDARY OUTCOMES:
Relapse rate | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Thomas, MD, FRCP(C), Principal Investigator — DermResearch @ 888 Inc.
Locations (1):
- Derm Research @ 888 Inc, Vancouver, British Columbia, Canada